CLINICAL TRIAL: NCT02784171
Title: A Phase II/III Randomized Study of Pembrolizumab in Patients With Advanced Malignant Pleural Mesothelioma
Brief Title: Pembrolizumab in Patients With Advanced Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: National Cancer Institute, Naples (Other); Merck Sharp & Dohme LLC (Industry); Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I227; 2016-002286-60 (EudraCT Number); IFCT-1901 (Other: Intergroupe Francophone de Cancerologie Thoracique)
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Cisplatin; Pemetrexed; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A - Cisplatin/Pemetrexed (Active Comparator): Pemetrexed 500 mg/m2 IV Day 1 every 21 days for 6 cycles Cisplatin 75 mg/m2 IV Day 1 every 21 days for 6 cycles
  Interventions: Drug: Cisplatin; Drug: Pemetrexed
- Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Active Comparator): Pembrolizumab 200 mg* IV Day 1 over 30 min every 21 days for a total of 2 years Pemetrexed 500 mg/m2 IV Day 1 every 21 days for 6 cycles Cisplatin 75 mg/m2 IV Day 1 every 21 days for 6 cycles
  Interventions: Drug: Cisplatin; Drug: Pemetrexed; Drug: Pembrolizumab
- Arm C - Pembrolizumab (Phase II only) (Active Comparator): Pembrolizumab 200 mg* IV 30 min Day 1 every 21 days for a total of 2 years
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Cisplatin
  Arms: Arm A - Cisplatin/Pemetrexed; Arm B - Cisplatin/Pemetrexed/Pembrolizumab
Drug: Pemetrexed
  Arms: Arm A - Cisplatin/Pemetrexed; Arm B - Cisplatin/Pemetrexed/Pembrolizumab
Drug: Pembrolizumab
  Arms: Arm B - Cisplatin/Pemetrexed/Pembrolizumab; Arm C - Pembrolizumab (Phase II only)

SUMMARY:
Pembrolizumab is a new type of drug for mesothelioma (immunotherapy). Laboratory tests show that this drug works by helping improve the body's immune response to help fight cancer. Pembrolizumab may help the immune system to recognize cancer cells and slow down the growth and/or spreading of cancer.

DETAILED DESCRIPTION:
The purpose of this study is to find out what effects a new drug, pembrolizumab has on this type of cancer and if it can offer better results than standard pemetrexed and platinum-based chemotherapy alone. This study will also look at side effects and how the treatments impact quality of life

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignant pleural mesothelioma. Patients must be eligible to receive standard chemotherapy with pemetrexed and cisplatin and have no contraindications to standard chemotherapy.
* Patients must have unresectable advanced and/or metastatic disease, incurable by standard therapies.
* All patients must have a cellular tumour block from their primary or metastatic tumour available and consent to release the block/recently cut slides for correlative analyses (See Section 11.0) and the centre/pathologist must have agreed to the submission of the specimen(s).
* Presence of radiologically documented disease. At least one site of disease must be unidimensionally measurable as follows:

  * CT scan (with slice thickness of ≤ 5 mm): ≥ 10 mm --> longest diameter
  * Physical exam (using calipers): ≥ 10 mm
  * Lymph nodes by CT scan ≥ 15 mm --> measured in short axis
* All radiology studies must be performed within 21 days prior to registration (exception: within 28 days if negative).
* Age ≥ 18 years.
* ECOG performance status 0 or 1.

Previous Therapy

Cytotoxic Chemotherapy:

* Patients must not have received prior chemotherapy for any stage of advanced/metastatic disease.
* Patients who received previous (neo)adjuvant cisplatin-based systemic chemotherapy must have received the last dose of chemotherapy at least 12 months before registration. Please contact CCTG PRIOR to randomization for such patients.

Other Anti-Cancer Therapy:

* Patients may not have received targeted small molecule therapy, immunotherapies and viral therapies, biologic therapies and angiogenesis inhibitors for advanced/metastatic disease, or any prior immunotherapy for any stage of disease.

Radiation:

* Patients may have had prior radiation therapy, but NOT to the thorax unless clear disease progression has been demonstrated and confirmed with CCTG. A minimum of 28 days must have elapsed between the end of radiotherapy and registration onto the study. Radiation must have involved < 30% of functioning bone marrow and there must be measurable disease outside the previously irradiated area (patients whose sole site of disease (for example pleural rind) is in a previously irradiated area are ineligible UNLESS there is evidence of progression, or new lesions have been documented, in the irradiated field). Please contact CCTG PRIOR to randomization if the patient has received prior thoracic radiation. Patients must have recovered from any acute toxic effects from radiation prior to registration.

Previous Surgery:

* Previous major surgery is permitted provided that it has been at least 28 days prior to patient registration and that wound healing has occurred.
* Lab Requirements:

  * Absolute neutrophils ≥ 1.5 x 10^9/L
  * Platelets ≥ 100 x 10^9/L
  * Hemoglobin ≥ 90 g/L
  * Bilirubin ≤ 1.5 x ULN (upper limit of normal)
  * AST and ALT ≤ 2.5 x ULN
  * Serum creatinine < 1.25 x ULN or Creatinine clearance ≥ 50 mL/min
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements.
* Patients must be accessible for treatment, response assessment and follow-up. Patients registered on this trial must be treated and followed at the participating centre.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient randomization.
* Women/men of childbearing potential must have agreed to use two highly effective contraceptive methods during the study and for six months after discontinuation.
* Patient must be able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires.

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (at doses more than 10 mg prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first and any dose of trial treatment.
* Has active autoimmune disease that has required systemic treatment in the past 3 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs) or history of allogeneic transplantation. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Must not have received a live vaccine within 30 days of planned start of study therapy.
* Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction including cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects) or who have had unstable angina congestive heart failure or myocardial infarction within the previous year. Patients with a significant cardiac history, this includes hypertension, even if controlled, should have a LVEF ≥ 50%.
* Patients with a history of other malignancies unless having undergone curative therapy (i.e. resection, radiation, etc) and do not require concurrent anticancer therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab or any of the other chemotherapy agents.
* Concurrent treatment with other investigational drugs or anti0cancer therapy.
* Patients with serious illness or medical condition that would not permit the patient to be managed according to the protocol including, but not limited to:

  * History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements.
  * Active infection requiring systemic therapy; (including any patient known to have active hepatitis B, hepatitis C or human immunodeficiency virus (HIV) [note: testing in asymptomatic patients is not required] or tuberculosis).
  * Known history of, or any evidence of active, non-infectious pneumonitis.
  * Any other medical conditions that might be aggravated by treatment.
  * Serious or non-healing wound, ulcer, or bone fracture.
* Patients with evidence of interstitial lung disease.
* Patients with severe/uncontrollable tumor pain that requires radiation prior to starting on systemic therapy.
* Pregnant or lactating women. (N.B.: All women of childbearing potential must have a negative pregnancy test within 72 hours prior to registration).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quincy Chu, Study Chair — Cross Cancer Institute, Edmonton Alberta Canada; Francesco Perrone, Study Chair — National Cancer Institute of Naples, Italy; Laurent Greillier Marseille, Study Chair — Hopital Nord, France
Locations (57):
- Canada (13):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University, Montreal, Quebec
  - University Institute of Cardiology and, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- France (25):
  - AP-HP Hopital Tenon, Paris, Cedex 20
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy, Cedex
  - CHU Dupuytren, Limoges, FR
  - Hopital du Scorff, Lorient, FR
  - Lyon URCOT, Pierre-Bénite, FR
  - CHU Rennes - Hopital Pontchaillou, Rennes, FR
  - Institut Gustave-Roussy, Villejuif, FR
  - CHRU de Tours - Hopital Bretonneau, Tours, Tours Cedex 9
  - CHU - Angers, Angers
  - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Boulogne - Ambroise Pare, Boulogne
  - Caen - CHU, Caen
  - Clermont-Ferrand - CHU, Clermont-Ferrand
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Centre Hospitalier du Mans, Le Mans
  - Lille - Hopital Calmette, Lille
  - Marseille - Hopital Nord, Marseille
  - Montpellier
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre Rene Gauducheau, Nantes
  - Hopital Bichat, Paris
  - Nouvel Hopital Civil Hopitaux, Strasbourg
  - CHITS Toulon Sainte Musse, Toulon
  - Hopital Larrey, Toulouse
- Italy (19):
  - Oncologia SS Antonio e Biagio Alessandria, Alessandria, AL
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino, AV
  - IRCCS Ospedale Oncologico Giovanni Paolo II, Bari, BA
  - Oncologia Medica Humanitas Gavazzeni Bergamo, Bergamo, BG
  - Azienda Ospedaliera Garibaldi Nesima, Catania, CT
  - Instituto Clinico Humanitas, Rozzano (MI), Lombardy
  - Oncologia Medica IRCCS Arcispedale Maria, Reggio Emilia, RE
  - Istituti Fisioterapici Ospitalieri IFO Istituto, Rome, RM
  - PO A Perrino ASL Brindisi - UOC Oncologia Medica, Brindisi
  - AOU Policlinico Vittorio Emanuele UOC di Oncologia, Catania
  - U.O. di Oncologia Ospedale Villa Scassi, Genova
  - Intstituto Scientifico Romangnolo, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - U.O.C. di Oncologia U.L.S.S. 13, Mirano
  - Azienda Ospedaliera di Rilievo Nazionale, Napoli
  - Dott. Fortunato Ciardiello,Cattedra Oncologia Medica, Napoli
  - U.O.S.D. Day Hospital Oncologico-Pneumologico, Napoli
  - Unita Sperimentazioni Cliniche Istituto per lo, Napoli
  - Azienda USL di Piacenza, Ospedale Gugliemimo Salieto, Piacenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chu Q, Perrone F, Greillier L, Tu W, Piccirillo MC, Grosso F, Lo Russo G, Florescu M, Mencoboni M, Morabito A, Cecere FL, Ceresoli GL, Dawe DE, Zucali PA, Pagano M, Goffin JR, Sanchez ML, Gridelli C, Zalcman G, Quantin X, Westeel V, Gargiulo P, Delfanti S, Tu D, Lee CW, Leighl N, Sederias J, Brown-Walker P, Luo Y, Lantuejoul S, Tsao MS, Scherpereel A, Bradbury P, Laurie SA, Seymour L. Pembrolizumab plus chemotherapy versus chemotherapy in untreated advanced pleural mesothelioma in Canada, Italy, and France: a phase 3, open-label, randomised controlled trial. Lancet. 2023 Dec 16;402(10419):2295-2306. doi: 10.1016/S0140-6736(23)01613-6. Epub 2023 Nov 3. PMID 37931632
- [Derived] Uprety D. CheckMate 743: A Glimmer of Hope for Malignant Pleural Mesothelioma. Clin Lung Cancer. 2021 Mar;22(2):71-73. doi: 10.1016/j.cllc.2020.11.009. Epub 2020 Dec 2. No abstract available. PMID 33358660

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - Cisplatin/Pemetrexed (Phase II); Arm A - Cisplatin/Pemetrexed (Phase III): Pemetrexed 500 mg/m2 IV Day 1 every 21 days for 6 cycles Cisplatin 75 mg/m2 IV Day 1 every 21 days for 6 cycles
  Cisplatin
  Pemetrexed
- Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Phase II); Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Phase III): Pembrolizumab 200 mg* IV Day 1 over 30 min every 21 days for a total of 2 years Pemetrexed 500 mg/m2 IV Day 1 every 21 days for 6 cycles Cisplatin 75 mg/m2 IV Day 1 every 21 days for 6 cycles
  Cisplatin
  Pemetrexed
  Pembrolizumab
- Arm C - Pembrolizumab (Phase II Only): Pembrolizumab 200 mg* IV 30 min Day 1 every 21 days for a total of 2 years
  Pembrolizumab
Period: Overall Study
Arm/Group | Arm A - Cisplatin/Pemetrexed (Phase II) | Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Phase II) | Arm C - Pembrolizumab (Phase II Only) | Arm A - Cisplatin/Pemetrexed (Phase III) | Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Phase III)
Started | 21 | 19 | 40 | 218 | 222
Completed | 21 | 19 | 40 | 218 | 222
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Phase III): Pembrolizumab 200 mg* IV Day 1 over 30 min every 21 days for a total of 2 years Pemetrexed 500 mg/m2 IV Day 1 every 21 days for 6 cycles Cisplatin 75 mg/m2 IV Day 1 every 21 days for 6 cycles
- Total: Total of all reporting groups
Arm/Group | Arm A - Cisplatin/Pemetrexed (Phase II) | Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Phase II) | Arm C - Pembrolizumab (Phase II Only) | Arm A - Cisplatin/Pemetrexed (Phase III) | Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Phase III) | Total
Number analyzed (Participants) | 21 | 19 | 40 | 218 | 222 | 520
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 14 | 61 | 42 | 129
  >=65 years | 16 | 12 | 26 | 157 | 180 | 391
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68.5 [65.4 to 74.2] | 69 [63.6 to 73] | 69.1 [62 to 73.8] | 70.8 [63.5 to 75.7] | 70.8 [66.4 to 75.3] | 70.5 [65.1 to 75.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 50 | 57 | 116
  Male | 19 | 16 | 36 | 168 | 165 | 404
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1
  White | 20 | 18 | 38 | 172 | 175 | 423
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 45 | 46 | 93
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 11 | 22 | 67 | 70 | 185
  Italy | 6 | 8 | 18 | 106 | 106 | 244
  France | 0 | 0 | 0 | 45 | 46 | 91

OUTCOME MEASURES:

1. Primary Outcome: Phase II: Progression Free Survival Measured as Time From Randomization to First Observation of Objective Disease Relapse or Progression
Description: PFS was calculated for all randomized patients from the day of randomization until the first observation of disease progression (date of objective relapse or progression of Relapse/Progression Report) or death due to any cause (recorded in Date/Cause of Death Section of Death Report).
Time Frame: PFS was monitored continuously, with assessments every 6 weeks for 3 visits, then every 12 weeks, 4 weeks post-discontinuation, every 12 weeks until progression, and every 24 weeks until death, over an average of 16.2 months.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A - Cisplatin/Pemetrexed: Pemetrexed 500 mg/m2 IV Day 1 every 21 days for 6 cycles Cisplatin 75 mg/m2 IV Day 1 every 21 days for 6 cycles
  Cisplatin
  Pemetrexed
- Arm B - Cisplatin/Pemetrexed/Pembrolizumab: Pembrolizumab 200 mg* IV Day 1 over 30 min every 21 days for a total of 2 years Pemetrexed 500 mg/m2 IV Day 1 every 21 days for 6 cycles Cisplatin 75 mg/m2 IV Day 1 every 21 days for 6 cycles
  Cisplatin
  Pemetrexed
  Pembrolizumab
Arm/Group | Arm A - Cisplatin/Pemetrexed | Arm B - Cisplatin/Pemetrexed/Pembrolizumab | Arm C - Pembrolizumab (Phase II Only)
Number analyzed (Participants) | 21 | 19 | 40
months | 6.7 [2.7 to 8.4] | 6.8 [3.9 to 15] | 5.26 [2.8 to 11.8]

2. Primary Outcome: Phase III: Overall Survival Defined as Time From Randomization to the Date of Death From Any Cause
Description: Overall survival was defined as time from the day of randomization to death for patients died. For patients still alive at time of data-cutoff for analysis, it was censored at the last day the patients were known alive as the last of all dates .
Time Frame: Survival was monitored continuously throughout the study and during follow-up. Patients were evaluated for each cycle, 4 weeks after discontinuation, every 12 weeks until progression, and then every 24 weeks until death, an average of 16.2 months.
Population: Intention to treat population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Cisplatin/Pemetrexed | Arm B - Cisplatin/Pemetrexed/Pembrolizumab
Number analyzed (Participants) | 218 | 222
months | 16.13 [13.08 to 18.17] | 17.28 [14.36 to 21.29]
Statistical Analysis 1: Comparison: Arm A - Cisplatin/Pemetrexed vs Arm B - Cisplatin/Pemetrexed/Pembrolizumab; Test type: Superiority; p = 0.0372, Log Rank

3. Secondary Outcome: Phase III: Progression Free Survival Measured as Time From Randomization to First Observation of Objective Disease Relapse or Progression
Description: PFS was calculated for all randomized patients from the day of randomization until the first observation of disease progression (date of objective relapse or progression of Relapse/Progression Report) or death due to any cause (recorded in Date/Cause of Death Section of Death Report). The primary analysis for PFS was based on the progression evaluated in this study using mesothelioma-modified RECIST (mRECIST) conducted by blinded independent review (BICR).
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Cisplatin/Pemetrexed | Arm B - Cisplatin/Pemetrexed/Pembrolizumab
Number analyzed (Participants) | 218 | 222
months | 7.16 [6.83 to 7.69] | 7.13 [6.93 to 8.12]

4. Secondary Outcome: Phase III: Objective Response Rate
Description: Objective response rate was defined as the proportion of patients with best objective response being complete response (CR) or partial response (PR).
Time Frame: Response was monitored continuously, with assessments every 6 weeks for 3 visits, then every 12 weeks, 4 weeks post-discontinuation, every 12 weeks until progression, and every 24 weeks until death, over an average of 16.2 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Cisplatin/Pemetrexed | Arm B - Cisplatin/Pemetrexed/Pembrolizumab
Number analyzed (Participants) | 218 | 222
Participants | 83 | 138

ADVERSE EVENTS:
Time Frame: Adverse events were monitored continuously throughout the study and during follow-up. Patients were evaluated before each cycle, 4 weeks after discontinuation, every 12 weeks until progression, and then every 24 weeks until death, an average of 16.2 months.
Arm/Group | Arm A - Cisplatin/Pemetrexed (Phase II) | Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Phase II) | Arm C - Pembrolizumab (Phase II Only) | Arm A - Cisplatin/Pemetrexed (Phase III) | Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Phase III)
All-Cause Mortality (participants affected / at risk) | 21/21 | 14/19 | 38/40 | 175/218 | 167/222
Serious Adverse Events (participants affected / at risk) | 8/21 | 10/19 | 13/40 | 38/218 | 92/222
Other Adverse Events (participants affected / at risk) | 20/21 | 18/19 | 38/40 | 200/218 | 217/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Cisplatin/Pemetrexed (Phase II) (N=21) | Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Phase II) (N=19) | Arm C - Pembrolizumab (Phase II Only) (N=40) | Arm A - Cisplatin/Pemetrexed (Phase III) (N=218) | Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Phase III) (N=222)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 7
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 11
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 3
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 2
Cardiac disorders - Other specify (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 3 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 2
Blurred vision (Eye disorders) | 0 | 0 | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 3
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 3
Death NOS (General disorders) | 0 | 0 | 1 | 0 | 1
Edema limbs (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 3 | 2
Fever (General disorders) | 0 | 0 | 0 | 2 | 6
General disorders and administration site conditions - Other specify (General disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Sudden death NOS (General disorders) | 0 | 1 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 1
Immune system disorders - Other specify (Immune system disorders) | 0 | 0 | 0 | 0 | 4
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 3
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infections and infestations - Other specify (Infections and infestations) | 0 | 0 | 0 | 3 | 3
Lung infection (Infections and infestations) | 0 | 1 | 1 | 5 | 9
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 7
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 4
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 4
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1
GGT increased (Investigations) | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 1 | 0 | 1 | 5
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Neoplasms benign malignant and unspecified (incl cysts and polyps) - Other specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2 | 3 | 7
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Myelitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0 | 1 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 3
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 4 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 8
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory thoracic and mediastinal disorders - Other specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Social circumstances - Other specify (Social circumstances) | 0 | 0 | 0 | 0 | 2
Hematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 5 | 5
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Cisplatin/Pemetrexed (Phase II) (N=21) | Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Phase II) (N=19) | Arm C - Pembrolizumab (Phase II Only) (N=40) | Arm A - Cisplatin/Pemetrexed (Phase III) (N=218) | Arm B - Cisplatin/Pemetrexed/Pembrolizumab (Phase III) (N=222)
Blood and lymphatic system disorders - Other specify (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 3
Atrial flutter (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac disorders - Other specify (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 2 | 6
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ear and labyrinth disorders - Other specify (Ear and labyrinth disorders) | 0 | 1 | 1 | 2 | 4
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 2
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 2 | 0 | 13 | 10
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 4 | 1 | 0 | 14 | 18
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 2 | 4
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 1 | 2 | 3
Hypothyroidism (Endocrine disorders) | 0 | 3 | 6 | 4 | 19
Blurred vision (Eye disorders) | 0 | 2 | 3 | 4 | 13
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 17 | 13
Dry eye (Eye disorders) | 0 | 0 | 0 | 12 | 9
Eye disorders - Other specify (Eye disorders) | 0 | 0 | 0 | 8 | 10
Eye pain (Eye disorders) | 1 | 0 | 0 | 1 | 3
Flashing lights (Eye disorders) | 0 | 0 | 0 | 0 | 1
Floaters (Eye disorders) | 0 | 0 | 1 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 1 | 1
Watering eyes (Eye disorders) | 3 | 2 | 0 | 14 | 29
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 2 | 12 | 33
Anal mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Anal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 3 | 4 | 4
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 5
Constipation (Gastrointestinal disorders) | 11 | 8 | 14 | 55 | 82
Diarrhea (Gastrointestinal disorders) | 4 | 6 | 9 | 30 | 67
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 3 | 5 | 12
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 4 | 14 | 19
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 3 | 6 | 11
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Esophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 4 | 0 | 8 | 6
Gastrointestinal disorders - Other specify (Gastrointestinal disorders) | 0 | 2 | 2 | 5 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 5
Mucositis oral (Gastrointestinal disorders) | 7 | 7 | 1 | 37 | 47
Nausea (Gastrointestinal disorders) | 13 | 13 | 9 | 99 | 120
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 3
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 7 | 1 | 35 | 57
Chills (General disorders) | 1 | 1 | 1 | 2 | 8
Edema face (General disorders) | 0 | 1 | 0 | 5 | 5
Edema limbs (General disorders) | 0 | 3 | 5 | 19 | 26
Edema trunk (General disorders) | 1 | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 17 | 14 | 24 | 141 | 153
Fever (General disorders) | 3 | 4 | 4 | 18 | 50
Flu like symptoms (General disorders) | 0 | 5 | 6 | 6 | 15
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0
General disorders and administration site conditions - Other specify (General disorders) | 0 | 0 | 0 | 0 | 5
Infusion related reaction (General disorders) | 1 | 1 | 0 | 2 | 8
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 1
Irritability (General disorders) | 0 | 0 | 0 | 1 | 0
Localized edema (General disorders) | 0 | 0 | 0 | 4 | 4
Malaise (General disorders) | 0 | 0 | 0 | 3 | 1
Neck edema (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 6 | 8 | 40 | 51
Pain (General disorders) | 2 | 1 | 6 | 13 | 14
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 1 | 1 | 1 | 3
Immune system disorders - Other specify (Immune system disorders) | 0 | 0 | 0 | 0 | 5
Bladder infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Bronchial infection (Infections and infestations) | 0 | 2 | 1 | 1 | 2
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gum infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Infections and infestations - Other specify (Infections and infestations) | 0 | 2 | 0 | 5 | 12
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lip infection (Infections and infestations) | 0 | 1 | 0 | 1 | 2
Lung infection (Infections and infestations) | 1 | 1 | 1 | 8 | 13
Mucosal infection (Infections and infestations) | 1 | 1 | 4 | 7 | 9
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Papulopustular rash (Infections and infestations) | 0 | 1 | 2 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Penile infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Pleural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 3
Skin infection (Infections and infestations) | 0 | 1 | 1 | 1 | 5
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Upper respiratory infection (Infections and infestations) | 0 | 3 | 1 | 2 | 11
Urethral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 4 | 5 | 15
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 7
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 5 | 10
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 3
Injury poisoning and procedural complications - Other specify (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 3
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 8 | 6 | 10 | 55 | 65
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 7 | 13
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 7 | 3 | 28
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 8 | 28 | 36
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 4 | 11
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 8 | 28 | 28
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1 | 7
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 5 | 7
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 5
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3 | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 1 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 8 | 12 | 22
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Neoplasms benign malignant and unspecified (incl cysts and polyps) - Other specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2 | 13 | 16
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Concentration impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 3
Dizziness (Nervous system disorders) | 3 | 1 | 3 | 15 | 24
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Dysesthesia (Nervous system disorders) | 0 | 0 | 0 | 3 | 2
Dysgeusia (Nervous system disorders) | 4 | 2 | 2 | 29 | 27
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 3 | 5 | 12 | 21
Ischemia cerebrovascular (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 2 | 5
Movements involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Myelitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Nervous system disorders - Other specify (Nervous system disorders) | 1 | 1 | 0 | 2 | 2
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 2 | 4
Paresthesia (Nervous system disorders) | 1 | 1 | 2 | 12 | 21
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1 | 0 | 1 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 5 | 4 | 19 | 31
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Sinus pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 0 | 0 | 2 | 1
Spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 1 | 0 | 0 | 3 | 4
Tremor (Nervous system disorders) | 0 | 0 | 0 | 4 | 7
Agitation (Psychiatric disorders) | 1 | 1 | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 6 | 3 | 2 | 12 | 16
Confusion (Psychiatric disorders) | 1 | 1 | 2 | 5 | 3
Depression (Psychiatric disorders) | 2 | 2 | 0 | 4 | 10
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 2 | 4 | 7 | 16 | 32
Mania (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 5
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 4
Hematuria (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 5
Renal and urinary disorders - Other specify (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 5
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 2 | 6 | 9
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 4
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 6
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 3 | 5 | 13
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 1 | 4 | 2
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Genital edema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Gynecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 4
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 2 | 1 | 2
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Reproductive system and breast disorders - Other specify (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 6 | 12
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 11 | 13 | 55 | 70
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 11 | 22 | 93 | 118
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 7 | 13
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 5 | 12
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 3 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 12 | 16
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 10
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 3 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 5 | 11 | 12
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Respiratory thoracic and mediastinal disorders - Other specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 9
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 4 | 7
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 6 | 12
Body odor (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 7 | 3 | 17
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 1
Fat atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 4 | 9
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 5 | 12 | 40
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 3 | 4 | 7 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 5 | 7 | 18 | 37
Skin and subcutaneous tissue disorders - Other specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 14 | 27
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 4 | 3
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2
Surgical and medical procedures - Other specify (Surgical and medical procedures) | 0 | 0 | 1 | 2 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 5
Hematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 3
Hot flashes (Vascular disorders) | 1 | 0 | 1 | 4 | 6
Hypertension (Vascular disorders) | 0 | 2 | 1 | 7 | 10
Hypotension (Vascular disorders) | 1 | 0 | 2 | 9 | 6
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 2 | 1
Superficial thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 3
Thromboembolic event (Vascular disorders) | 3 | 1 | 2 | 16 | 26
Vascular disorders - Other specify (Vascular disorders) | 0 | 1 | 0 | 1 | 5
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT02784171/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT02784171/SAP_001.pdf